CLINICAL TRIAL: NCT01977651
Title: A Multicenter, Single-arm, Open-label, Postmarketing Safety Study to Evaluate the Risk of Seizure Among Subjects With Metastatic Castration-Resistant Prostate Cancer (mCRPC) Treated With Enzalutamide Who Are at Potential Increased Risk of Seizure
Brief Title: A Study to Evaluate the Potential Increased Risk of Seizures Among Metastatic Castration-Resistant Prostate Cancer (mCRPC) Patients Treated With Enzalutamide
Acronym: UPWARD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Collaborators: Medivation LLC, a wholly owned subsidiary of Pfizer Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9785-CL-0403; 2013-003022-92 (EudraCT Number); U1111-1157-0224 (Registry Identifier: World Health Organization (WHO))
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Results first posted 2020-12-09 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Castration-resistant Prostate Cancer (mCRPC)
Keywords: enzalutamide; Xtandi; seizure; Central Nervous System; MDV3100; metastatic castration-resistant prostate cancer (mCRPC)
MeSH Terms: conditions — Seizures | interventions — enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Enzalutamide 160 mg (Experimental): Participants received 160 mg of enzalutamide orally once a day, for 4 months. At the end of the 4-month treatment period, participants who were assessed as deriving benefit from enzalutamide treatment continued in the extension period. The total study drug treatment duration for the extended period depended on individual clinical benefit. If a participant experienced a Grade 3 or higher toxicity that was attributed to enzalutamide and could not be ameliorated by the use of adequate medical intervention, treatment with enzalutamide was allowed to be interrupted for 1 week or until the toxicity grade improved to Grade 2 or lower severity. Subsequently, enzalutamide was restarted at the original dose 160 mg per day or a reduced dose 120 or 80 mg per day in consultation with the medical monitor.
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Enzalutamide — Participants received 4 capsules (40 mg each) of enzalutamide orally once a day, for a total daily dose of 160 mg. Treatment was given with or without food and as close as possible to the same time each day.
  Other Names: Xtandi; MDV3100

SUMMARY:
The objective of this study was to evaluate the incidence of seizures and monitor the safety of enzalutamide treatment in participants with metastatic castration-resistant prostate cancer (mCRPC) known to have risk factor(s) for seizure.

DETAILED DESCRIPTION:
This was a multicenter, single-arm, open-label, postmarketing safety study to evaluate the risk of seizure among patients with mCRPC treated with enzalutamide who were at potential increased risk of seizure.

Participants who met all inclusion and none of the exclusion criteria were enrolled into the study and participated in a 4-month treatment period, during which once daily dosing of enzalutamide (160 mg/day) occurred. At the end of the 4-month treatment period, participants who were assessed as deriving benefit from enzalutamide treatment were allowed to continue in the extension period where participants continued to receive enzalutamide until 1 of the following criteria was met:

1. The participant experienced bone disease progression per Prostate Cancer Working Group 2 (PCWG2) guidelines or soft tissue disease progression per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1
2. The participant initiated treatment with another anticancer therapy or, in the opinion of the investigator, continued dosing would have led to undue risk to the patient
3. The participant met a discontinuation criterion
4. The sponsor terminated the study

Participants who continued to receive clinical benefit from treatment with enzalutamide and did not meet any discontinuation criteria may have transitioned to an open label roll-over extension study upon approval of the study protocol at the institution where they were receiving treatment.

Participants who did not continue in the extension period or who met a discontinuation criterion were discontinued from enzalutamide therapy and completed a follow-up visit 30 days from the last dose of enzalutamide or prior to the initiation of another anticancer therapy, whichever occurred first.

For participants who continued on treatment after the 12-month extension period, data collection was limited to dosing information, concomitant medications, and all adverse events (AEs) including serious adverse events (SAEs).

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically confirmed metastatic adenocarcinoma of the prostate.
* Subject has ongoing androgen deprivation therapy with a Gonadotropin-releasing hormone (GnRH) analogue (agonist or antagonist) or bilateral orchiectomy (i.e., surgical or medical castration).
* Subject has disease progression by at least one of the following:

  1. Prostate-Specific Antigen (PSA) progression defined by a minimum of 2 rising PSA levels with an interval of at least 1 week between each draw;
  2. Bone disease progression as defined by Prostate Cancer Working Group 2 guidelines (at least 2 new lesions) on bone scan; or
  3. Soft tissue disease progression as defined by RECIST 1.1
* For subjects who have not had an orchiectomy, there must be a plan to maintain effective GnRH-analogue therapy for the duration of the study.
* Subject must have failed at least one course of androgen deprivation therapy (ADT), i.e., treatment with GnRH analogues.
* Subject has an Eastern Cooperative Oncology Group (ECOG) performance status of 0-2.
* Subject has been evaluated by a local neurologist prior to study entry who has determined the subject has at least one risk factor for seizure including:

  1. past history of seizure due to any cause except a single febrile seizure in childhood. Patients with a history of seizures should not have had a seizure within 12 months of Screening and must have had no anticonvulsants for 12 months prior to Screening,
  2. history of cerebrovascular accident (CVA) or transient ischemic attack (TIA),
  3. history of traumatic brain or head injury with loss of consciousness
  4. unexplained loss of consciousness within the last 12 months,
  5. presence of a space occupying lesion in the brain including previously treated brain metastasis(es) or primary central nervous system (CNS) tumor,
  6. history of arteriovenous malformations of the brain,
  7. history of brain infection (i.e., abscess, meningitis, or encephalitis),
  8. current use of medication that may lower seizure threshold
  9. presence of Alzheimer's disease, meningioma, leptomeningeal disease from prostate cancer.
* Subject is able to swallow the study drug and comply with study requirements.
* Subject agrees not to participate in another interventional study while on treatment.
* Male subject and his female partner who is of childbearing potential must use two acceptable methods of birth control (one of which must include a condom as a barrier method of contraception) starting at Screening and continuing throughout the study period and for 3 months after final study drug administration.

  1. Two acceptable forms of birth control include:
  1. Condom (barrier method of contraception), AND
  2. One of the following acceptable forms of contraception is required:

     1. Established use of oral, injected or implanted hormonal methods of contraception.
     2. Placement of an intrauterine device (IUD) or intrauterine system (IUS).
     3. Barrier methods of contraception: Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository).
     4. Vasectomy or surgical castration at least 6 months prior to Screening.
* Male subject must use a condom, if having sex with a pregnant woman.
* Male subject must not donate sperm starting at Screening and throughout the study period and for at least 3 months after final drug administration.

Exclusion Criteria:

* Subject with a history of exposure to enzalutamide.
* Subject has severe concurrent disease, infection, or co-morbidity that, in the judgment of the Investigator, would make the subject inappropriate for enrollment.
* Subject is currently being treated with anti-epileptics.
* Subject has a history of seizure within the past 12 months of Screening as assessed by neurology examination and history.
* Subject with rapidly progressing visceral disease who has not received and is thought to be able to tolerate cytotoxic chemotherapy. (However, subject who has previously received cytotoxic chemotherapy is permitted).
* Subject has clinical signs suggestive of high or imminent risks for pathological fracture, spinal cord compression and/or cauda equina syndrome.
* Subject's absolute neutrophil count is < 1500/microliter (µL), platelet count is < 100,000/µL) or hemoglobin is < 5.6 millimoles(mmol)/liter (L) (9 grams (g)/deciliter (dL) at Screening.
* Subject's total bilirubin is ≥ 1.5 x upper limit of normal (ULN) (except for subjects with documented Gilbert's disease) or alanine aminotransferase (ALT) or aspartate aminotransferase (AST) is ≥ 2.5x upper limit of normal (ULN) at Screening.
* Subject's estimated creatinine clearance (Cer) is less than 30 milliliter (mL)/minute (min) by the Cockcroft and Gault formula (Creatinine Clearance (mL/min) = (140 - age)(weight (wt) kilogram (kg) / 72 x serum creatinine (milligram (mg)/100 mL) [Cockcroft, 1976] at Screening.
* Subject has uncontrolled hypertension as indicated by a resting systolic blood pressure > 160 millimeter of mercury (mmHg) or diastolic blood pressure > 100 millimeter of mercury (mmHg) at Screening.
* Subject has received an investigational agent within 4 weeks or 5 half lives whichever is longer prior to Day 1.
* Subject has shown a hypersensitivity reaction to the active pharmaceutical ingredient or any of the capsule components, including Labrasol, butylated hydroxyanisole, and butylated hydroxytoluene.

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2013-09-25 (Actual); Primary Completion 2016-02-01 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (76):
- United States (9):
  - Site US10005, Anchorage, Alaska
  - Site US10024, Detroit, Michigan
  - Site US10001, New York, New York
  - Site US10014, New York, New York
  - Site US10039, Syracuse, New York
  - Site US10026, The Bronx, New York
  - Site US10016, Durham, North Carolina
  - Site US10008, Dallas, Texas
  - Site US10025, Seattle, Washington
- Argentina (6):
  - Site AR54001, Berazategui, Buenos Aires
  - Site AR54006, Ciudad Autonoma de BuenosAires, Buenos Aires
  - Site AR54002, Buenos Aires, Buenos Aires F.D.
  - Site AR54003, Córdoba
  - Site AR54005, San Miguel de Tucumán
  - Site AR54004, Santa Fe
- Australia (7):
  - Site AU61012, Kogarah, New South Wales
  - Site AU61005, Randwick, New South Wales
  - Site AU61011, Sydney, New South Wales
  - Site AU61001, Tweed Heads, New South Wales
  - Site AU61002, Nambour, Queensland
  - Site AU61007, Adelaide, South Australia
  - Site AU61004, Ballarat, Victoria
- Belgium (3):
  - Site BE32004, Anderlecht
  - Site BE32001, Kortrijk
  - Site BE32003, Liège
- Canada (5):
  - Site CA15005, Abbotsford, British Columbia
  - Site CA15014, Halifax, Nova Scotia
  - Site CA15004, Brampton, Ontario
  - Site CA15010, Scarborough Village, Ontario
  - Site CA15001, Québec, Quebec
- Chile (4):
  - Site CL56001, Temuco, Región de la Araucanía
  - Site CL56004, Santiago
  - Site CL56002, Temuco
  - Site CL56003, Viña del Mar
- Czechia (2):
  - Site CZ42004, Prague
  - Site CZ42002, Prague
- Finland (3):
  - Site FI35803, Helsinki
  - Site FI35801, Oulu
  - Site FI35802, Tampere
- France (3):
  - Site FR33002, Lyon
  - Site FR33004, Rouen
  - Site FR33005, Suresnes
- Germany (3):
  - Site DE49009, Nürtingen, Baden-Wurttemberg
  - Site DE49003, Berlin
  - Site DE49001, Münster
- Site HU36002, Sopron, Győr-Moson-Sopron, Hungary
- Israel (8):
  - Site IL97202, Kfar Saba, Central District
  - Site IL97203, Beersheba
  - Site IL97201, Be’er Ya‘aqov
  - Site IL97205, Haifa
  - Site IL97204, Jerusalem
  - Site IL97208, Nahariya
  - Site IL97206, Petah Tikva
  - Site IL97207, Ramat Gan
- Italy (4):
  - Site IT39005, Meldola, Emilia-Romagna
  - Site IT39001, Cremona, Lombardy
  - Site IT39002, Arezzo
  - Site IT39003, Roma
- Site NZ64001, Hamilton, New Zealand
- Site SG65002, Singapore, Singapore
- South Korea (5):
  - Site KR82006, Seongnam-si, Gyeonggi-do
  - Site KR82007, Seoul
  - Site KR82003, Seoul
  - Site KR82001, Seoul
  - Site KR82004, Seoul
- Spain (6):
  - Site ES34007, L'Hospitalet de Llobregat, Barcelona
  - Site ES34005, Sabadell, Barcelona
  - Site ES34001, Pamplona, Navarre
  - Site ES34003, Barcelona
  - Site ES34004, Barcelona
  - Site ES34006, Madrid
- Sweden (2):
  - Site SE46001, Gothenburg
  - Site SE46002, Örebro
- Taiwan (2):
  - Site TW88601, Kaohsiung City
  - Site TW88603, Taipei
- Site GB44002, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to results on the Astellas Clinical Study Results website. — https://astellasclinicalstudyresults.com/study.aspx?ID=349

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study enrolled male participants with histologically-confirmed metastatic adenocarcinoma of prostate with ongoing androgen deprivation therapy with a gonadotropin-releasing hormone (GnRH) analogue (agonist or antagonist) or a prior orchiectomy. Participants were evaluated by a neurologist who determined they had at least 1 risk factor for seizure.
Pre-assignment Details: Participants who met all inclusion and none of the exclusion criteria were enrolled in the study, completing a 4-month treatment period. Participants who benefited from the treatment were allowed to continue in the extension period. A total 424 participants were enrolled and 423 participants received the study drug.
Period: 4 Month Treatment Period
Arm/Group | Enzalutamide 160 mg
Started | 423
Completed | 322
Not Completed | 101
Not completed — Adverse Event | 34
Not completed — Death | 3
Not completed — Progressive Disease | 43
Not completed — Withdrawal by Subject | 17
Not completed — Physician Decision | 4
Period: 1 Year Extension Period
Arm/Group | Enzalutamide 160 mg
Started | 287 (Participants who benefited from enzalutamide treatment continued in the 1 year extension period)
Completed | 157
Not Completed | 130
Not completed — Adverse Event | 14
Not completed — Death | 10
Not completed — Lost to Follow-up | 2
Not completed — Progressive Disease | 86
Not completed — Withdrawal by Subject | 11
Not completed — Physician Decision | 6
Not completed — Miscellaneous | 1
Period: Post 1 Year Extension Period
Arm/Group | Enzalutamide 160 mg
Started | 145 (Participants who benefited from enzalutamide treatment continued in the post 1 year extension period)
Completed | 1
Not Completed | 144
Not completed — Adverse Event | 5
Not completed — Death | 13
Not completed — Progressive Disease | 60
Not completed — Withdrawal by Subject | 13
Not completed — Physician Decision | 4
Not completed — Miscellaneous | 49

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) consisted of all participants who took at least 1 dose of study drug and for whom any data was reported after first dose of study drug.
Groups:
- Enzalutamide 160 mg: Participants received 160 mg of enzalutamide orally once a day, for 4 months.
Arm/Group | Enzalutamide 160 mg
Number analyzed (Participants) | 423
Age, Continuous [Mean (Standard Deviation); unit: Years] | 73.2 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 423
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  WHITE | 381
  BLACK OR AFRICAN AMERICAN | 9
  ASIAN | 25
  NATIVE HAWAIIAN OR OTHER PACIFIC ISLANDER | 1
  NO DATA | 3
  OTHER | 4
Ethnicity [Count of Participants; unit: Participants]
  NOT HISPANIC OR LATINO | 331
  HISPANIC OR LATINO | 89
  NO DATA | 3
Eastern Cooperative Oncology Group (ECOG) At Study Entry [Number; unit: participants] — ECOG performance status is a scale used to measure disease progression and impact on daily activities. Scores range from 0 to 5, with grade 0- signifying fully active participant, grade 1-restricted in physically strenuous activity; grade 2 - ambulatory and capable of all self-care, unable to work; grade 3- capable of only limited self-care, confined to bed more than 50% of waking hours; grade 4-completely disabled and grade 5- dead.
  participants
    Grade 0 | 188
    Grade 1 | 190
    Grade 2 | 45

OUTCOME MEASURES:

1. Primary Outcome: The Percentage of Evaluable Participants With at Least One Confirmed Seizure as Adjudicated by the Independent Adjudication Committee (IAC)
Description: Percentage of evaluable participants with at least one confirmed seizure as adjudicated by the IAC during the first 4 months of treatment were reported.
Time Frame: Day 1 up to week 17 (end of 4-month treatment period)
Population: The seizure risk evaluation set (SRES) consisted of all participants with a confirmed seizure during the 4-month treatment period of the study or who completed at least 3 months (75 percent [%]) of the planned treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Enzalutamide 160 mg
Number analyzed (Participants) | 366
percentage of participants | 1.1 [0.3 to 2.8]

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (approximately 52 months)
Arm/Group | Enzalutamide 160 mg
All-Cause Mortality (participants affected / at risk) | 62/423
Serious Adverse Events (participants affected / at risk) | 193/423
Other Adverse Events (participants affected / at risk) | 318/423
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide 160 mg (N=423)
Anaemia (Blood and lymphatic system disorders) | 9 (11)
Anaemia of malignant disease (Blood and lymphatic system disorders) | 1 (1)
Aplastic anaemia (Blood and lymphatic system disorders) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 2 (2)
Angina pectoris (Cardiac disorders) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 4 (5)
Atrial flutter (Cardiac disorders) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure (Cardiac disorders) | 4 (5)
Cardiac failure chronic (Cardiac disorders) | 1 (2)
Cardiac failure congestive (Cardiac disorders) | 3 (4)
Cardiogenic shock (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 5 (6)
Right ventricular failure (Cardiac disorders) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (3)
Hypoacusis (Ear and labyrinth disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Blindness (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 6 (6)
Colonic obstruction (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (3)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 2 (3)
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 4 (5)
Proctalgia (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 7 (8)
Asthenia (General disorders) | 3 (4)
Chest pain (General disorders) | 1 (1)
Death (General disorders) | 1 (1)
Device leakage (General disorders) | 1 (1)
Drug ineffective (General disorders) | 1 (1)
Fatigue (General disorders) | 3 (3)
Gait disturbance (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 10 (18)
Glassy eyes (General disorders) | 1 (1)
Multi-organ failure (General disorders) | 1 (1)
Pain (General disorders) | 5 (6)
Performance status decreased (General disorders) | 1 (1)
Pyrexia (General disorders) | 8 (10)
Spinal pain (General disorders) | 1 (1)
Sudden cardiac death (General disorders) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 1 (2)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1)
Anal abscess (Infections and infestations) | 1 (1)
Appendicitis (Infections and infestations) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1)
Bronchopneumonia (Infections and infestations) | 2 (3)
Candiduria (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Clostridium difficile colitis (Infections and infestations) | 1 (1)
Corona virus infection (Infections and infestations) | 1 (1)
Cystitis (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (2)
Erysipelas (Infections and infestations) | 1 (1)
Escherichia urinary tract infection (Infections and infestations) | 2 (2)
Localised infection (Infections and infestations) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (2)
Pneumonia (Infections and infestations) | 13 (16)
Pyelonephritis (Infections and infestations) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 3 (3)
Respiratory tract infection (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 4 (4)
Spinal cord infection (Infections and infestations) | 1 (1)
Streptococcal urinary tract infection (Infections and infestations) | 1 (1)
Tracheobronchitis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (4)
Urinary tract infection bacterial (Infections and infestations) | 3 (3)
Urinary tract infection enterococcal (Infections and infestations) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 2 (2)
Urosepsis (Infections and infestations) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 10 (10)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 4 (4)
Hip fracture (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 2 (4)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 2 (2)
Upper limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Urostomy complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
C-reactive protein increased (Investigations) | 1 (1)
Cystoscopy (Investigations) | 1 (2)
Haemoglobin decreased (Investigations) | 1 (1)
Prostatic specific antigen increased (Investigations) | 2 (2)
Cachexia (Metabolism and nutrition disorders) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 5 (5)
Failure to thrive (Metabolism and nutrition disorders) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (4)
Hypophagia (Metabolism and nutrition disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 8 (8)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 3 (3)
Pubic pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign neoplasm of ureter (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cholangiocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 34 (39)
Metastases to liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Metastases to lymph nodes (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Altered state of consciousness (Nervous system disorders) | 1 (1)
Brain stem stroke (Nervous system disorders) | 1 (1)
Carotid artery stenosis (Nervous system disorders) | 1 (2)
Central nervous system haemorrhage (Nervous system disorders) | 1 (1)
Cerebral artery occlusion (Nervous system disorders) | 1 (1)
Cerebral artery stenosis (Nervous system disorders) | 1 (3)
Cerebral haemorrhage (Nervous system disorders) | 2 (3)
Cerebral infarction (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Cognitive disorder (Nervous system disorders) | 1 (1)
Convulsion (Nervous system disorders) | 8 (10)
Diplegia (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Haemorrhagic stroke (Nervous system disorders) | 1 (2)
IIIrd nerve paralysis (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 2 (2)
Loss of consciousness (Nervous system disorders) | 2 (2)
Nerve root compression (Nervous system disorders) | 1 (1)
Normal pressure hydrocephalus (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 7 (8)
Syncope (Nervous system disorders) | 5 (5)
Transient global amnesia (Nervous system disorders) | 2 (3)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Agitation (Psychiatric disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 10 (10)
Delirium (Psychiatric disorders) | 2 (2)
Disorientation (Psychiatric disorders) | 1 (1)
Fear of falling (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Panic attack (Psychiatric disorders) | 1 (1)
Paranoia (Psychiatric disorders) | 1 (1)
Anuria (Renal and urinary disorders) | 1 (2)
Bladder dilatation (Renal and urinary disorders) | 1 (1)
Dysuria (Renal and urinary disorders) | 4 (4)
Haematuria (Renal and urinary disorders) | 8 (12)
Hydronephrosis (Renal and urinary disorders) | 2 (2)
Nephritic syndrome (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 4 (4)
Renal failure acute (Renal and urinary disorders) | 4 (5)
Urethral stenosis (Renal and urinary disorders) | 2 (3)
Urinary bladder haemorrhage (Renal and urinary disorders) | 1 (2)
Urinary retention (Renal and urinary disorders) | 5 (7)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 (6)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 4 (6)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bladder lesion excision (Surgical and medical procedures) | 1 (1)
Internal fixation of fracture (Surgical and medical procedures) | 1 (1)
Joint arthroplasty (Surgical and medical procedures) | 1 (1)
Aortic aneurysm (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Hypertension (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enzalutamide 160 mg (N=423)
Anaemia (Blood and lymphatic system disorders) | 53 (82)
Constipation (Gastrointestinal disorders) | 46 (50)
Diarrhoea (Gastrointestinal disorders) | 43 (54)
Nausea (Gastrointestinal disorders) | 55 (65)
Vomiting (Gastrointestinal disorders) | 24 (29)
Asthenia (General disorders) | 86 (113)
Fatigue (General disorders) | 92 (120)
Oedema peripheral (General disorders) | 33 (39)
Pain (General disorders) | 23 (28)
Fall (Injury, poisoning and procedural complications) | 24 (31)
Weight decreased (Investigations) | 26 (27)
Decreased appetite (Metabolism and nutrition disorders) | 77 (92)
Arthralgia (Musculoskeletal and connective tissue disorders) | 47 (56)
Back pain (Musculoskeletal and connective tissue disorders) | 68 (82)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 22 (24)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 27 (33)
Headache (Nervous system disorders) | 25 (26)
Insomnia (Psychiatric disorders) | 27 (34)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 33 (37)
Hot flush (Vascular disorders) | 24 (26)
Hypertension (Vascular disorders) | 31 (36)

LIMITATIONS AND CAVEATS:
After completing the extension period participants who were assessed to benefit from enzalutamide completed their treatment in another Astellas study, 9785-CL-0123 (NCT02960022).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2016-10-20): https://cdn.clinicaltrials.gov/large-docs/51/NCT01977651/Prot_000.pdf
  • Statistical Analysis Plan (2014-03-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT01977651/SAP_001.pdf